CLINICAL TRIAL: NCT03337672
Title: Comparison of Dexmedetomidine and Midazolam for Prevention of Emergence Delirium in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunah Cho, MD (Other)
Responsible Party: Sponsor-Investigator, Eunah Cho, MD, Clinical Assistant Professor, Kangbuk Samsung Hospital
Organization: Kangbuk Samsung Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017-04-038-001
Record Dates: First submitted 2017-11-01; First posted 2017-11-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Tonsillitis
MeSH Terms: conditions — Tonsillitis | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Subjects who receive dexmedetomidine for prevention of emergence delirium
  Interventions: Drug: Dexmedetomidine
- Midazolam group (Active Comparator): Subjects who receive midazolam for prevention of emergence delirium
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous dexmedetomidine 0.3mcg/kg is slowly infused at 5 minutes before the end of surgery
  Arms: Dexmedetomidine group
Drug: Midazolam — Intravenous dexmedetomidine 0.03mg/kg is slowly infused at 5 minutes before the end of surgery
  Arms: Midazolam group

SUMMARY:
Emergence delirium is a common complication in children after anesthesia. The incidence of emergence delirium is reported upto 50%. Prevention of emergence delirium in children is important not only for the patient safety but also for the satisfaction of the parents. Midazolam is the most commonly used medications for prevention of emergence delirium. However, it might lead to delayed awakening from anesthesia and respiratory depression. In this study, the investigators will evaluate whether dexmedetomidine can be effectively and safely administered for prevention of emergence delirium in children compared to midazolam.

DETAILED DESCRIPTION:
In this study, seventy patients scheduled for elective tonsillectomy aged from 24 months to 12 years old Anesthesiologists physical status (ASA) class 1 and 2 will be enrolled. The sample size was calculated based on the former study with a type 1 error estimate of 0.05 at 80% power. The proportion in dexmedetomidine group (group D) was assumed to be 0.4 and the proportion in midazolam group (group M) was 0.1. Considering the drop-out rate of 10%, seventy patients in total were needed.The patients will randomly be allocated into the group D or the group M. The group D will receive dexmedetomidine0.3mcg/kg mixed with 0.9% normal saline, 10mL in total. The group M will receive 0.03mg/kg of midazolam mixed with 0.9% normal saline, 10mL in total. Randomization and drug administration will be done by a single anesthesiologist. Assessment of the patient will be done by another anesthesiologist blinded by the group. Five minutes before the end of the surgery, the study drug will be slowly infused for 5 minutes. In the postanesthesia circuit unit (PACU), presence of emergence delirium will be assessed. The emergence delirium will be assessed by the four-point agitation scale. (1 = calm, 2 = not calm but gould be easily calmed, 3 = not easily calmed, moderately agitated or restless, and 4 = combative, exited or disoriented.) Patients with score 3 and 4 will be diagnosed as emergence delirium and treated with intravenous fentanyl 1mcg/kg. Severity of emergence delirium will be assessed with the pediatric anesthesia emergence delirium scale after 10 mins on arrival of PACU. Pain wil be scored by 5-point scale (0 = no pain, 5 = severe pain ever). Time from discontinuation of anesthetic gas to extubate will be recorded. The data will be compared between the groups by the independent t-test or Mann-Whitney test for the continuous variables. Chi-square test or Fisher's exact test will be used for the categorial variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective tonsillectomy under general anesthesia
* American society of anesthesiologist physical status 1,2
* aged from 24 months to 12 years old
* obtaining written informed consent

Exclusion Criteria:

* known history of allergy to dexmedetomidine or midazolam
* renal impairment
* hepatic impairment
* long QT syndrome
* developmental disorder
* congenital disorder
* neurologic disorder
* psychogenic disorder

Ages: 24 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Presence of Emergence Delirium (ED) | 0 minute, 5 minutes, 10 minutes, 15 minutes and 20 minutes after arrival at the PACU
  During the PACU stay, the patients will be assessed whether the emergence delirium (ED) occurred. It is defined as ED, if the highest score is more than 3 points after five time point measurements by the four-point agitation scale (1=calm, 2=not calm but easily calmed, 3=not easily calmed, moderately agitated, and 4=combative, excited, disoriented). The five time points are the 0 minute, 5 minutes, 10 minutes, 15 minutes and 20 minutes after arrival at the PACU.

SECONDARY OUTCOMES:
Severity of Emergence Delirium | 10 minutes after arrival at the PACU
  Patients will be scored using the pediatric anesthesia emergence delirium scale. This consists of 5 criteria, each of which is pointed from 0 to 5 according to the severity. Total score stands for the delirium severity.
Emergence time | 3 minutes after extubation
  Time from the discontinuation of the anesthetic gas to extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Eunah Cho, M.D., Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea